CLINICAL TRIAL: NCT02441738
Title: Hybrid Thoracoscopic Surgical and Transvenous Catheter Ablation Versus Transvenous Catheter Ablation in Persistent and Longstanding Persistent Atrial Fibrillation
Brief Title: Hybrid Versus Catheter Ablation in Persistent AF
Acronym: HARTCAP-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL.52951.068.16
Record Dates: First submitted 2015-05-04; First posted 2015-05-12 (Estimated); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Hybrid Ablation; Catheter Ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hybrid Ablation (Active Comparator): Epicardial surgical ablation performed thoracoscopically with occlusion/removal of the LAA combined with percutaneous endocardial ablation (one-stage).
  Interventions: Procedure: Hybrid Ablation
- Catheter Ablation (Active Comparator): Percutaneous endocardial catheter ablation, with optional repeated catheter ablation(s).
  Interventions: Procedure: Catheter Ablation

INTERVENTIONS:
Procedure: Hybrid Ablation — The procedure will be performed following standard of care guidelines.
  Arms: Hybrid Ablation
Procedure: Catheter Ablation — The procedure will be performed following standard of care guidelines.
  Arms: Catheter Ablation

SUMMARY:
Atrial fibrillation (AF) is the most common cardiac arrhythmia with a lifetime risk of developing AF of 1 in 4 people aged over 40. Besides hemodynamic compromises stroke remains the most feared complication of AF with an increase in risk by 5-fold.

Catheter ablation has evolved as a standardized treatment option in paroxysmal AF. Due to the advanced electrical and structural remodeling the single procedural results of catheter ablation for persistent and longstanding persistent AF are rather disappointing without a proven superiority of any applied strategy compared to others. However, repeated catheter ablation can achieve better results. The surgical (epicardial) approach seems to be more effective, though still a significant amount of failures exist. Checking the epicardial ablation lines and if necessary making additional endocardial lines (which is a hybrid ablation) is expected to be most efficacious in avoiding lesion gaps and providing the most complete lesion set.

The study objective of this pilot trial is to compare the safety and efficacy of catheter ablation within 6 months versus a hybrid ablation consisting of endoscopic epicardial surgery combined with endocardial catheter ablation (performed one-stage) in preventing the recurrence of atrial fibrillation (AF) in symptomatic, drug refractory patients with persistent or longstanding persistent atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Known with a history of symptomatic persistent AF or longstanding persistent atrial fibrillation,
* Refractory to or intolerant of at least one antiarrhythmic drug class I or III,
* At least 18 years of age,
* Mentally able and willing to give informed consent.

Exclusion Criteria:

* Previous ablation procedure,
* Longstanding persistent AF > 3 years,
* Paroxysmal atrial fibrillation. Successful cardioversion within 48 hours of onset of the arrhythmia will be also considered paroxysmal. In patients with paroxysmal and persistent AF, the dominant pattern should be taken to categorize,
* Atrial fibrillation secondary to electrolyte imbalance, thyroid disease, or other reversible or non-cardiovascular cause,
* Presence of left atrial appendage (LAA) thrombus,
* Left atrial size ≥ 60mm (PLAX-view on TEE),
* Left ventricular ejection fraction < 40%,
* In need for other cardiac surgery then AF treatment within 12 months,
* Intolerance to heparin and warfarin,
* Unable to undergo TEE,
* Sick-sinus-syndrome
* Mitral valve insufficiency > Iº
* Carotic stenosis > 80%,
* Active infection or sepsis,
* Pleural adhesions,
* Elevated hemi diaphragm
* Significant pulmonary dysfunction as assessed by preoperative lung testing,
* Chronic obstructive pulmonary disease with a FEV1 or VC < 50% predicted
* History of cerebrovascular accident (CVA) or transient ischemic attack (TIA),
* History of blood clotting abnormalities,
* History of thoracic radiation,
* History of pericarditis,
* History of cardiac tamponade,
* History of thoracotomy or cardiac surgery,
* Body-mass-index > 40,
* Pregnancy,
* Life expectancy less than 12 months,
* Participation in any other clinical study involving an investigational drug or device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-10-31 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Freedom from any AT off antiarrhythmic drugs class I or III lasting > 5 minutes after the blanking period, evaluated by any ECG-tracing and 7-day holter. | 12 Months
Major complications during follow-up | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Pison, MD, PhD, Principal Investigator — Maastricht University Medical Center; Mark La Meir, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] van der Heijden CAJ, Weberndorfer V, Vroomen M, Luermans JG, Chaldoupi SM, Bidar E, Vernooy K, Maessen JG, Pison L, van Kuijk SMJ, La Meir M, Crijns HJGM, Maesen B. Hybrid Ablation Versus Repeated Catheter Ablation in Persistent Atrial Fibrillation: A Randomized Controlled Trial. JACC Clin Electrophysiol. 2023 Jul;9(7 Pt 2):1013-1023. doi: 10.1016/j.jacep.2022.12.011. Epub 2023 Jan 18. PMID 36752455
- [Derived] Vroomen M, La Meir M, Maesen B, Luermans JGL, Vernooy K, Essers B, de Greef BTA, Maessen JG, Crijns HJ, Pison L. Hybrid thoracoscopic surgical and transvenous catheter ablation versus transvenous catheter ablation in persistent and longstanding persistent atrial fibrillation (HARTCAP-AF): study protocol for a randomized trial. Trials. 2019 Jun 20;20(1):370. doi: 10.1186/s13063-019-3365-9. PMID 31221218